CLINICAL TRIAL: NCT01898624
Title: Specified Drug Use-results Survey of Betanis Tablets in OAB Patients With Coexisting Glaucoma
Brief Title: Specified Drug Use-results Survey of Betanis Tablets
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: BE0004
Record Dates: First submitted 2013-07-10; First posted 2013-07-12 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Overactive Bladder
Keywords: mirabegron; Overactive Bladder; Betanis®; glaucoma
MeSH Terms: conditions — Urinary Bladder, Overactive; Glaucoma | interventions — mirabegron

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Betanis group: mirabegron treated group
  Interventions: Drug: mirabegron

INTERVENTIONS:
Drug: mirabegron — oral
  Other Names: Betanis; YM178

SUMMARY:
To investigate the effects of mirabegron on the symptoms of glaucoma in overactive bladder (OAB) patients with coexisting glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as OAB and treated with mirabegron
* diagnosed as glaucoma (including normal tension glaucoma)
* having intraocular pressure measurement conducted more than twice within six months before the start of the mirabegron treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: OAB patients with coexisting glaucoma treated with mirabegron
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2012-12-04 (Actual); Primary Completion 2018-01-10 (Actual); Study Completion 2018-01-10 (Actual)

PRIMARY OUTCOMES:
The occurrence of ocular adverse events such as increased intraocular pressure and worsening of glaucoma | 12 weeks

SECONDARY OUTCOMES:
Changes in OABSS (Over Active Bladder Symptoms Score) | Baseline and 12 weeks of treatment
  OABSS is judged by investigator

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma Inc
Locations (7):
- Japan (7):
  - Chugoku
  - Chūbu
  - Kansai
  - Kanto
  - Kyushu
  - Shikoku
  - Tōhoku

IPD SHARING:
Plan to Share IPD: Undecided